CLINICAL TRIAL: NCT04704518
Title: Phase IV Clinical Study to Evaluate the Efficacy of Lagricel® Ofteno PF Compared to Thealoz® Duo for Corneal Re-epithelialization After Photorefractive Keratectomy (PRK)
Brief Title: Phase IV Study to Evaluate the Efficacy of Lagricel® Ofteno PF Compared to Thealoz® Duo After Photorefractive Keratectomy (PRK)
Acronym: PRO-037
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOPH037-0120/IV
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-12

CONDITIONS: Photorefractive Keratectomy; Corneal De-epithelialization
MeSH Terms: interventions — Trehalose

STUDY DESIGN:
Intervention Model Description: Comparative, controlled, parallel group, open, randomized multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1; Lagricel® Ofteno PF (Experimental): Lagricel® Ofteno PF, multidose presentation (sodium hyaluronate 0.4%) Ophthalmic Solution. One drop QID, both eyes (OU) for 14 days.
  Interventions: Drug: Sodium Hyaluronate Ophthalmic 0.4%
- Group 2; Thealoz® Duo (Active Comparator): Thealoz® Duo, (trehalose 3%/sodium hyaluronate 0.15%). Ophthalmic Solution. One drop QID, both eyes (OU) for 14 days.
  Interventions: Drug: Trehalose 3% / Sodium Hyaluronate Ophthalmic 0.15%

INTERVENTIONS:
Drug: Sodium Hyaluronate Ophthalmic 0.4% — Topical ophthalmic administration of one drop of Lagricel® Ofteno PF QID.
  Other Names: Lagricel® Ofteno PF; PRO-037
  Arms: Group 1; Lagricel® Ofteno PF
Drug: Trehalose 3% / Sodium Hyaluronate Ophthalmic 0.15% — Topical ophthalmic administration of one drop of Thealoz® Duo QID.
  Other Names: Thealoz® Duo
  Arms: Group 2; Thealoz® Duo

SUMMARY:
Phase IV comparative, controlled, parallel group, open, randomized multicenter study to evaluate the efficacy of Lagricel® Ofteno PF Compared to Thealoz® Duo. Primary outcome measure is the time of corneal re-epithelialization after PRK surgery. Intervention includes administration of one of the experimental products quater per die (QID) for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 and ≤ 45 years old
* Being on PRK postoperative day 1 (right eye will be evaluated for efficacy)
* Presenting a PRK surgical corneal ablation surface of 5.5 to 6.0 mm
* PRK corneal output ≤ 60 µm
* Preoperative refraction of -1.0 to -4.5 D of myopia or myopic astigmatism (in this case, the sum of both values with a spherical equivalent no greater than -4.5 D)
* Being capable of voluntarily grant a signed informed consent.
* Being willing and able to meet the requirements of the study such as attending programmed visits, treatment plan and other study procedures.
* Being willing and able to modify the required lifestyle activities.
* Women in child-bearing age must assure the continuation (start ≥ 30 days prior to informed consent signing) of a hormonal contraceptive method or intrauterine device (IUD) during the study.

Exclusion Criteria:

* Having suffered any complications during and after PRK surgical procedure previous to inclusion in the study.
* Use of mitomycin during PRK
* Being subjected to PRK retreatment of previous history of any other kind of refractive surgery.
* Pregnancy, breastfeeding or planning to become pregnant during the time of the study
* Having participated in clinical trials within 30 days prior to signing this study's informed consent form.
* Having participated previously in this study.
* Diagnosis of any of the following:

  * Allergic, viral or bacterial conjunctivitis
  * Dry eye
  * Anterior blepharitis
  * Parasite infestation of ocular structures (Demodex, for example)
  * Previous history of ocular herpes
  * Previous history of ocular inflammation (such as uveitis)
  * Corneal or conjunctival ulcers
  * Glaucoma
* Previous history of drug addiction within the last 2 years previous to signing this study's informed consent form.
* Having a previous history of any ophthalmological surgical procedure, within the last 3 months prior to the informed consent signing date.
* Previous history of any medical affliction, acute or chronic (such as Diabetes Mellitus type I/II, autoimmune diseases or HIV), that according to the investigator may increase either the risk to the patient for participating in this study or the risk of interference of the accurate interpretation of results.
* Use of medications (such as retinoic acid) that according to the investigator's criteria may increase either the risk to the patient for participating in this study or the risk of interference of the accurate interpretation of results.
* Known hypersensitivity to any of the components of the products used in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2022-09-03 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Changes in corneal re-epithelialization (time) | Days: 1 (baseline visit), 2 (±1) (first follow-up visit), 3 (±1) (second follow-up visit), 7 (±1) (third follow-up visit)
  Corneal re-epithelialization will be evaluated through direct observation and photographic recording after application of fluorescein stain. After instillation of a drop of topical anesthetic (tetracaine 0.5%) a fluorescein strip will be applied on the inferior cul de sac while the patient looks upward. Using a slit lamp with magnification of 6x and 16x photographs (at least 6 images for each magnification) will be obtained.
Incidence of adverse events | Day: 15 (±1) (final visit)
  Presence/absence adverse events, defined as the appearance of any unfavorable reaction in a patient participating in a clinical investigation in which any pharmaceutical product is being administered, regardless of the causal attribution.
Change in Best Corrected Visual Acuity (BCVA) | Days: 1 (baseline visit), 2 (±1) (first follow-up visit), 3 (±1) (second follow-up visit), 7 (±1) (third follow-up visit) and 15 (±1) (final visit)
  With the patient's best possible refractive correction, visual acuity will be evaluated through the Snellen chart. Its notation (fraction or decimal) is described as the distance from the chart at which the test is performed, divided by the distance at which a letter equals vertically 5 minutes of arc.

SECONDARY OUTCOMES:
Changes in Ocular Comfort Index | Days: 7 (±1) (third follow-up visit) and 15 (±1) (final visit)
  Ocular Comfort Index (OCI) Questionnaire will be used for evaluation of tolerability through incidence and severity of dry eye symptoms in a scale from 0 to 100. Greater scores mean a worse outcome.
Pain perception | Days: 1 (baseline visit), 2 (±1) (first follow-up visit), 3 (±1) (second follow-up visit), 7 (±1) (third follow-up visit) and 15 (±1) (final visit)
  Through a questionnaire, patients will be directly questioned about presence and severity of pain and associated symptoms. The scale will be as follows for severity: absent (0), very mild (1), mild (2), moderate (3) and severe (4); and for frequency: never (0), almost never (1), 50% of the time (2), almost all the time (3) and all the time (4).

CONTACTS AND LOCATIONS:
Locations (1):
- Aris Vision Institute de Guadalajara, S. C., Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No